CLINICAL TRIAL: NCT04954287
Title: A Phase 1 Open-Label, Dose-Ranging Trial to Evaluate the Safety and Immunogenicity of Intranasal Parainfluenza Virus Type 5- SARS CoV-2 S Vaccine (CVXGA1) in Healthy Adults Aged 18 to 55 Years and Adolescents Aged 12 to 17 Years
Brief Title: Phase 1 Study of Intranasal PIV5 COVID-19 Vaccine Expressing SARS-CoV-2 Spike Protein in Healthy Adults and Adolescents
Acronym: CVXGA1-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CyanVac LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CVXGA1-001
Record Dates: First submitted 2021-06-30; First posted 2021-07-08 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Covid19
Keywords: Intranasal Vaccine; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — CVXGA1 COVID-19 vaccine

STUDY DESIGN:
Intervention Model Description: Progression will be by dose escalation (low dose to high dose) in healthy adults aged 18 to 55 years (N=up to 60), with approximately 12 months' follow-up. Safety data from sentinel subjects (4) will be assessed by a safety monitoring committee (SMC) if halting rules are met for 1) vaccine administration to the remaining subjects within the group, 2) progression from the low dose (1 x 106 PFU) group to the high dose (1 x 107 PFU) groups (without or with prior receipt of COVID vaccine), and 3) progression from the high dose adult group (18 to 55 years) with prior receipt of COVID vaccine to the adolescent (12-17 years) group (N= up to 20) with prior receipt of COVID-19 vaccine.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1, 1 x 10^6 PFU CVXGA1 in Ages 18-55 (Experimental): Group 1 (Young adults aged 18 to 55 years - CVXGA1- Low Dose, no prior COVID vaccine or infection)
  Interventions: Biological: CVXGA1 low dose
- Group 2, 1 x 10^7 PFU CVXGA1 in Ages 18-55 (Experimental): Group 2 (Young adults aged 18 to 55 years - CVXGA1- High Dose, no prior COVID vaccine, no prior COVID vaccine or infection allowed if occurring at least 5 months prior to enrollment)
  Interventions: Biological: CVXGA1 high dose
- Group 3, 1 x 10^7 PFU CVXGA1 in Ages 18-55 (Experimental): Group 3 (Young adults aged 18-55 years - CVXGA1 - High Dose, prior receipt of two or more doses of COVID mRNA vaccine (Pfizer Comirnaty® or Moderna Spikevax™) at least 5 months prior to study enrollment. Prior COVID infection allowed if occurring at least 5 months prior to study enrollment).
  Interventions: Biological: CVXGA1 high dose
- Group 4, 1 x 10^7 PFU CVXGA1 in Ages 12-17 (Experimental): Group 4 (Adolescents aged 12-17 years - CVXGA1 - High Dose, prior receipt of two or more doses of COVID mRNA vaccine (Pfizer Comirnaty® or Moderna Spikevax™) at least 5 months prior to study enrollment. Prior COVID infection allowed if occuring at least 5 months prior to study enrollment.
  Interventions: Biological: CVXGA1 high dose

INTERVENTIONS:
Biological: CVXGA1 low dose — see arm/group description
  Other Names: PIV5-SARS CoV-2 vaccine
  Arms: Group 1, 1 x 10^6 PFU CVXGA1 in Ages 18-55
Biological: CVXGA1 high dose — see arm/group description
  Other Names: PIV5-SARS CoV-2 vaccine
  Arms: Group 2, 1 x 10^7 PFU CVXGA1 in Ages 18-55; Group 3, 1 x 10^7 PFU CVXGA1 in Ages 18-55; Group 4, 1 x 10^7 PFU CVXGA1 in Ages 12-17

SUMMARY:
This Phase 1 trial is an open-label trial to evaluate the safety, reactogenicity and immunogenicity of two dosages (10^6 PFU and 10^7 PFU) of intranasal CVXGA1 administered as a single dose in healthy adults age 18-55 years and in adolescents age 12-17.

DETAILED DESCRIPTION:
This is an open-label, dose-ranging phase 1 trial of the PIV5 virus-vectored SARS CoV-2 S glycoprotein vaccine (CVXGA1) in healthy adults (males and nonpregnant females) 18 to 55 years of age that have not had a prior COVID vaccination (Groups 1 and 2), and in healthy adults 18 to 55 years of age (Groups 3) and adolescents 12-17 years of age (Group 4) who have received at least two doses of mRNA-based COVID vaccines (Pfizer Comirnaty® or Moderna Spikevax™) with the last dose at least 5 months prior to planned receipt of CVXGA1 study vaccine. The trial is designed to assess the safety, reactogenicity, and immunogenicity of a single dose of intranasal CVXGA1. Two dose levels will be assessed, CVXGA1-low lose (LD) at 106 plaque-forming units (PFU) (Group 1) and CVXGA1-high dose (HD) at 107 PFU (Groups 2, 3 and 4).

ELIGIBILITY:
Inclusion Criteria:

1. Provide informed consent and assent as applicable prior to initiation of any trial procedures.
2. Be able to understand and agrees to comply with planned trial procedures and be available for all trial visits.
3. Agrees to the collection of venous blood per protocol.
4. Healthy male or non-pregnant female between 12 and 55 years of age inclusive at time of enrollment who are not at high risk of SARS-CoV-2 exposure defined as individuals whose health status, profession, locations or circumstances put them at high risk of exposure to SARS-CoV-2 and COVID-19.
5. Body Mass Index (BMI) <40.0 kg/m2 (or < 35.0 kg/m2 if obesity-related health conditions are present) at screening. Subjects must weigh a minimum of 31 kg.
6. Women of childbearing potential* must agree to use or have practiced true abstinence** or use at least one acceptable primary form of contraception.***, **** Note: These criteria are applicable to females in a heterosexual relationship and child-bearing potential (i.e., the criteria do not apply to subjects in a same sex relationship).
7. Women of childbearing potential must have a negative urine or serum pregnancy test within 24 hours prior to vaccination.
8. Male subjects of childbearing potential*: use of condoms to ensure effective contraception with a female partner of childbearing potential from vaccination until 90 days after vaccination. If barrier methods are to be used, then double barrier methods of protection are required i.e. male condom with a cap, diaphragm or sponge with spermicide. *Biological males who are post-pubertal and considered fertile until permanently sterile by bilateral orchiectomy or vasectomy.
9. Male subjects agree to refrain from sperm donation from the time of vaccination until 90 days after vaccination.
10. Female subjects agree to refrain from egg donation from time of vaccination until 90 days after vaccination.
11. In good health.*
12. Oral temperature of 97.0°F (36.1°C) to less than 100.4° Fahrenheit (37.8° C).
13. Pulse is less than 100 beats per minute.
14. Systolic blood pressure (BP) is 85 to 150 mmHg, inclusive.
15. Diastolic blood pressure <95 mmHg, inclusive. Repeat blood pressure measurements are permitted.
16. Clinical screening laboratory evaluations (white blood cells (WBC) [total and differential counts], hemoglobin, platelets, alanine transaminase, aspartate transaminase, creatinine, alkaline phosphatase, total bilirubin, lipase, prothrombin time and partial thromboplastin time) are within acceptable normal reference ranges at the clinical laboratory being used. Alternatively, the clinical laboratory abnormalities grading scale noted in the FDA Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers enrolled in Preventive Vaccine Clinical Trials may be used.
17. Must agree to have samples stored for secondary research.
18. Agrees to adhere to pandemic public health guidance on preventing SARS-CoV-2 infection (e.g. wearing a mask, keeping physically distant, sheltering-in) throughout trial duration.
19. Must agree to refrain from donating blood or plasma during the trial (outside of this trial).
20. Seronegative to SARS-CoV-2 for subjects in Group 1, 2, and negative for SARS-CoV-2 by PCR at screening for all Groups.
21. For Groups 3 and 4 only, documented receipt of at least two-doses of COVID mRNA vaccine (any combination of Pfizer Comirnaty® and Moderna Spikevax™ vaccines) with the last dose at least 5 months prior to planned dosing of CVXGA1, and without receipt of any other COVID vaccines. In addition, subjects may not have had known COVID-19 infection in the 5 months prior to planned dosing of CVXGA1 study vaccine.

Exclusion Critera:

1. Positive pregnancy test either at screening or just prior to vaccine administration.
2. Female subject who is breastfeeding or plans to breastfeed from the time of the vaccination through 60 days after vaccination.
3. Anyone at high risk of severe COVID-19 disease as per current CDC guidance (< https://www.cdc.gov/coronavirus/2019-ncov/hcp/clinical-care/underlyingconditions.html>) or has any medical disease or condition that, in the opinion of the participating site PI or appropriate sub-investigator, precludes trial participation.* *Including acute, subacute, intermittent or chronic medical disease or condition that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this trial.
4. Presence of self-reported or medically documented significant medical or psychiatric condition(s).*
5. Has an acute illness*, as determined by the participating site PI or appropriate sub- investigator, with or without fever [oral temperature ≥ 38.0° Celsius (100.4° Fahrenheit)] within 72 hours of vaccination. *An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the participating site PI or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol.
6. Has a positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus (HIV) types 1 or 2 antibodies at screening.
7. Has participated in another investigational trial involving any investigational product (unlicensed vaccine, drug, biologic, device, blood product, or medication) within 60 days, or 5 half-lives, whichever is longer, before vaccine administration.
8. Currently enrolled in or plans to participate in another clinical trial with an investigational product (unlicensed vaccine, drug, biologic, device, blood product, or medication) that will be received during the trial-reporting period.
9. Has previously participated in an investigational trial of prophylaxis or treatment for SARS-CoV-2 infection or COVID-19 disease, except for Groups 3 and 4, who may have previously participated in investigational trials in which the subject received only the Pfizer Comirnaty® and/or Moderna Spikevax™ vaccines.
10. Has a history of hypersensitivity or severe allergic reaction (e.g., anaphylaxis, generalized urticaria, angioedema, other significant reaction) to any previous licensed or unlicensed vaccines.
11. Chronic use (more than 14 continuous days) of any medications that may be associated with impaired immune responsiveness.*
12. Anticipating the need for immunosuppressive treatment within the next 6 months.
13. Received immunoglobulins and/or any blood or blood products within the 4 months before vaccine administration or at any time during the trial.
14. Has any blood dyscrasias or significant disorder of coagulation.
15. Has any chronic liver disease, including fatty liver.
16. Has a history of alcohol abuse or other recreational drug (excluding cannabis) use within 6 months before vaccine administration.
17. Received or plans to receive a licensed, live vaccine within 4 weeks before or after vaccination.
18. Received or plans to receive a licensed, inactivated vaccine within 2 weeks before or after vaccination.
19. Prior receipt of a COVID-19 vaccine (except for prior doses of the Pfizer Comirnaty® and/or Moderna Spikevax™ vaccines in subjects enrolled in Groups 3 and 4), or planned receipt of a COVID-19 vaccine within the first 6 months after CVXGA1 study vaccine administration.
20. Close contact of anyone known to have SARS-CoV-2 infection within 14 days prior to CVXGA1 study vaccine administration.
21. History of COVID-19 diagnosis (positive test for antigen or PCR or antibody) at any time in the past (Group 1), or in the 5 months prior to CVXGA1 study vaccine administration (Groups 2, 3 and 4).
22. On current treatment with investigational agents for prophylaxis of COVID-19.
23. Plan to travel outside the United States (US) (continental US, Hawaii, and Alaska) from enrollment through 28 days after vaccination.
24. Reside in a nursing home or other skilled nursing facility or have a requirement for skilled nursing care.
25. Non-ambulatory.
26. For subjects of any age, individuals currently working with high risk of exposure to SARS-CoV-2.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2023-06-10 (Actual)

PRIMARY OUTCOMES:
Solicited Adverse Events | Day 1-8
  Frequencies and grades of solicited local and systemic AEs during a 7-day period after dosing
Unsolicited Adverse Events | Day 1-29
  Frequencies and grades of unsolicited AEs during the 28-day period after dosing

SECONDARY OUTCOMES:
Serum IgG titers to SARS-CoV-2 S protein | Day 29
  Geometric mean titer (GMT) of serum IgG titers specific to SARS-CoV-2 spike protein (S)
Percentage of subjects who seroconverted | Day 29
  Percentage of subjects who seroconverted, where seroconversion is defined as a ≥4-fold increase in titer from Baseline (Day 1) of serum IgG titers specific to SARS-CoV-2 spike protein (S)
Change in IgG titers to SARS-CoV-2 S protein | Day 29
  Geometric mean fold rise in titer from Baseline (GMFR) of serum IgG titers specific to SARS-CoV-2 spike protein (S)
Adverse Events within 30 min of dosing | Day 1
  Frequencies of AEs occurring within 30 minutes after dosing
Medically Attended Adverse Events | Day 1 - 181
  Frequencies of Medically Attended Adverse Events (MAAEs) from Day 1 to Day 181
Serious adverse events, new-onset chronic medical conditions, and adverse events of special interest | Day 1 to Day 366
  Frequencies of serious adverse events (SAEs), new-onset chronic medical condition (NOCMCs) and AEs of Special Interest (AESIs)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Spearman, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (4):
- United States (4):
  - Kentucky Pediatric/ Adult Research, Bardstown, Kentucky
  - University of Rochester Medical Center, Rochester, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Research Your Health, Plano, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD underlying the results reported in any published articles (text, tables, figures, appendices) will be shared.
Supporting Information: Study Protocol
Time Frame: 5 years, beginning as soon as possible (but no later than 12 months) after article publication
Access Criteria: Data will be made available to investigators and institutions upon request. Requests should be directed to the CyanVac authors of the publication(s).

REFERENCES:
- [Derived] Nakahashi-Ouchida R, Fujihashi K, Kurashima Y, Yuki Y, Kiyono H. Nasal vaccines: solutions for respiratory infectious diseases. Trends Mol Med. 2023 Feb;29(2):124-140. doi: 10.1016/j.molmed.2022.10.009. Epub 2022 Nov 23. PMID 36435633